CLINICAL TRIAL: NCT07345338
Title: Mainstreaming Genetic Testing for Non-Ischemic Cardiomyopathy in Western Canada: A Family-Centered and Genome-First Approach to a Common and Life-Threatening Cardiomyopathy
Brief Title: Mainstreaming Genetic Testing for Non-Ischemic Cardiomyopathy in Western Canada
Acronym: HOGI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Roston (Other)
Collaborators: Genome British Columbia (Industry); Genome Alberta (Other); University of Calgary (Other)
Responsible Party: Sponsor-Investigator, Thomas Roston, Principal Investigator, Cardiology Research UBC
Organization: Cardiology Research UBC (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: H25-02075
Record Dates: First submitted 2025-12-02; First posted 2026-01-15 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Nonischemic Cardiomyopathy; Dilated Cardiomyopathy (DCM)
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Intervention Model Description: Cluster randomized crossover trial with 4 sites (each province will have an intervention and control site; allocations will remain in place for the first 6 months - after 6 months, the sites switch allocations and begin enrolling new participants under these allocations).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mainstreamed Genetic Testing through Heart Function Clinics (Experimental): Mainstreamed genetic testing offered directly by the Heart Function Clinic cardiologist with video-based genetic counselling tools
  Interventions: Other: Health service delivery change
- Traditional Referral Pathway for Genetic Testing (No Intervention): Traditional referral pathway to a specialized cardiac genetics clinic

INTERVENTIONS:
Other: Health service delivery change — Genetic testing for patients with unexplained non-ischemic cardiomyopathy offered directly by cardiologists in Heart Function Clinics
  Arms: Mainstreamed Genetic Testing through Heart Function Clinics

SUMMARY:
Heart muscle disorders are a common cause of heart failure: a life-threatening condition that can cause dangerous abnormal heart rhythms (arrhythmia) and a buildup of fluid in the body (edema). In British Columbia (BC) and Alberta, patients with heart failure are cared for in specialized Heart Function Clinics (HFC). Providers in these clinics rapidly diagnose and treat heart failure because early treatment prevents death and disability. In some situations, particularly in young people, heart failure is caused by abnormalities in the genetic blueprint of the heart muscle - this is present at birth and passed down within families (i.e. hereditary). The investigators can diagnose this genetic abnormality by a simple blood or saliva test, which allows for better treatment of patients and diagnosis of family members to protect against heart failure and death. In BC and Alberta, people suspected of having this form of heart failure must be referred to highly specialized programs to receive genetic testing, as these healthcare systems currently do not offer genetic testing through HFCs. However, HFC providers are unaware or discouraged to refer patients because of very long waitlists of these programs. In this study, the investigators want to educate, enable, and empower HFC cardiologists to order genetic testing for heart failure. If such an intervention demonstrates success in this study, patients will no longer have to wait for up to 3 years to see a genetic specialist. Patients will be diagnosed and treated earlier, and their family members who might be in danger of having the condition can be informed more quickly. The investigators aim to leverage this study to encourage healthcare leadership to facilitate more timely access to genetic testing by showing the positive impact on health outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Clinical eligibility for non-ischemic cardiomyopathy/dilated cardiomyopathy (NICM/DCM) genetic testing, per existing clinical criteria in each respective province a. BC sites - presence of NICM/DCM with at least one of the following: i. Family history of NICM/DCM ii. Evidence of conduction disease iii. Arrhythmia (Ventricular or atrial) iv. Unexplained cardiomyopathy under 70 years v. Suggestive syndrome(s)

Alberta sites - Left ventricular ejection fraction of less than 50% and any degree of left or right ventricular dilation

Exclusion Criteria:

1. Previously known genetic result that explains NICM/DCM
2. Under age 18 years
3. Declines genetic testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Uptake of genetic testing for non-ischemic cardiomyopathy (NICM) | Through 12 months after first participant enrollment
  Proportion of eligible patients who complete clinical genetic testing for non-ischemic cardiomyopathy (NICM) following referral from a Heart Function Clinic.
Time to genotypic diagnosis | Up to 12 months after consent for genetic testing is provided.
  Time (in days) from the date informed consent for genetic testing is signed to the date genetic test results are returned.

SECONDARY OUTCOMES:
Proportion of participants with a change in clinical management following genetic test results | Up to 12 months after return of genetic test results
  Change in clinical management is defined as the initiation, discontinuation, or modification of at least one of the following, documented in the medical record after return of genetic test results:
  * Heart failure pharmacotherapy
  * Cardiac device therapy (e.g., implantable cardioverter-defibrillator [ICD], cardiac resynchronization therapy [CRT]) or transplantation
  * Referral to specialized services (e.g., inherited cardiomyopathy clinic, genetic counseling)
  * Pregnancy-related guidance or referral
  * Family cascade testing or screening recommendations
Patient-reported satisfaction, knowledge, and decision quality related to genetic testing | At 12 months after first participant enrollment
  Patient-reported outcomes assessed using a study-specific survey administered after receipt of information about genetic testing and discussion with a heart specialist. The survey includes:
  Knowledge items assessed using true/false/"I don't know" questions related to inherited heart disease and genetic testing
  Attitudinal items assessing views on genetic testing using 5-point Likert scales, where higher scores indicate more favorable views
  Experience and process items assessed using yes/no questions (e.g., whether sufficient time was provided)
  Decision satisfaction and decision quality items assessed using 5-point Likert scales ranging from strongly disagree (1) to strongly agree (5), with higher scores indicating greater satisfaction and alignment with personal values
Proportion of participants with a change to family screening recommendations following genetic test results | Up to 12 months after return of genetic test results
  Change in family screening recommendations is defined as any new, modified, or discontinued recommendation for screening of first- or second-degree relatives documented in the participant's medical record after return of genetic test results. This includes, but is not limited to:
  * Initiation of cascade genetic testing for relatives
  * Recommendations for cardiac imaging or surveillance in family members
  * Changes in age of screening initiation or screening interval
  * Determination that no family screening is recommended

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Roston, MD/PhD, Principal Investigator — University of British Columbia
Locations (4):
- Canada (4):
  - Peter Lougheed Centre Cardiac Function Clinic, Calgary, Alberta
  - Foothills Medical Centre Cardiac Function Clinic, Calgary, Alberta
  - Vancouver General Hospital Cardiac Function Clinic, Vancouver, British Columbia
  - St. Paul's Hospital Heart Function Clinic, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No